CLINICAL TRIAL: NCT01112891
Title: Vitamin D Dose-response Study Throughout Pregnancy and Lactation
Brief Title: Vitamin D in Pregnancy and Lactation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H09-01261; F08-03892 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Infant; Lactation; Dose-Response
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Vitamin D
- 2 (Experimental)
  Interventions: Drug: Vitamin D3
- 3 (Experimental)
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 10 ug/day Vitamin D as part of standard pre-natal vitamin supplement, taken from 18 weeks gestation to 6 months postpartum.
  Arms: 1
Drug: Vitamin D3 — 25 ug/day Vitamin D as part of standard pre-natal vitamin supplement, taken from 18 weeks gestation to 6 months postpartum.
  Arms: 2
Drug: Vitamin D — 50 ug/day Vitamin D as part of standard pre-natal vitamin supplement, taken from 18 weeks gestation to 6 months postpartum.
  Arms: 3

SUMMARY:
Background: Vitamin D is vital throughout pregnancy and lactation for both maternal and infant health. Health Canada recommends women take the AI of 5ug/day of vitamin D during pregnancy, however, it is unknown how much vitamin D is necessary to ensure both mother and baby reach a vitamin D serum concentration of 25OHD>75nmol/L.

DETAILED DESCRIPTION:
Purpose & Hypothesis: This project aims to determine maternal and infant responses vitamin D supplementation in pregnancy and lactation. It is hypothesized that the current AI of 5 μg of vitamin D will be inadequate for women and their infants in Canada to achieve optimal 25OHD concentrations (> 75nmol/L).

Methods: Healthy pregnant women between 18-42 years of age without history of pregnancy complications will be recruited for a double-blind, randomized, controlled trial where they will receive one of three different dosages of vitamin D (10, 25 and 50ug/day) as part of a standard prenatal vitamin. The study at 18 plus/minus 3 weeks gestation and will carry on throughout pregnancy and lactation. Mother and infant vitamin D levels in breast milk and blood will be measured at regular intervals. Skin colour will be measured via light reflectometry. Bone biomarkers such as plasma osteocalcin and urinary n-telopeptide will be assessed. Dietary vitamin D intake and sun exposure will be estimated using a food frequency and lifestyle questionnaire. Data will be analyzed using multiple regression analysis controlling for baseline values.

Expected Results & Conclusions: It is expected that greater vitamin D intakes (25, 50ug/day) will be necessary to raise maternal and infant serum concentrations to 25OHD>75nmol/L to avoid infant supplementation. This data will aid policy makers, mothers and healthcare workers in recommended and appropriate vitamin D dosage throughout pregnancy and lactation.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-42 years of age
* within 18 plus/minus 3 weeks gestation
* planning to breastfeed their infant
* a singleton pregnancy

Exclusion Criteria:

* Any co-morbid condition such pre-gestational diabetes, TB, cardiac or renal disease, HIV/AIDS, chronic hypertension, inflammatory bowel disease, autoimmune disease, liver disease, or epilepsy; conditions associated with vitamin D malabsorption: celiac disease, gastric bypass;
* History of previous adverse pregnancy outcome [preterm delivery <37; weeks GA, stillbirth, severe pre-eclampsia, eclampsia, HELLP syndrome (hemolytic anemia, elevated liver enzymes, and low platelet count)];
* Women will also be ineligible if they are taking more than 10 µg day supplemental vitamin D or drugs known to interfere with vitamin D metabolism (i.e corticosteroids).

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
25(OH)D Plasma Concentrations | 18 weeks gestation for mother
25(OH)D Plasma Concentrations | 28 weeks gestation for mother
25(OH)D Plasma Concentrations | 36 weeks gestation for mother
25(OH)D Plasma Concentrations | 16 weeks post-partum for mother & infant

CONTACTS AND LOCATIONS:
Overall Officials: Tim Green, Dr., Principal Investigator — University of British Columbia; Sheila M. Innis, Dr., Study Director — University of British Columbia; Michael R. Lyon, MD, Study Director — University of British Columbia; Antonia W. Shand, Dr, Study Director — University of British Columbia; Peter von Dadelszen, MD, Study Director — University of British Columbia; Russ Freisen, MSc, Study Chair — University of British Columbia; Kaitlin March, Study Chair — University of British Columbia; Tina Li, Study Chair — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Stamm RA, March KM, Karakochuk CD, Gray AR, Brown RC, Green TJ, Houghton LA. Lactating Canadian Women Consuming 1000 microg Folic Acid Daily Have High Circulating Serum Folic Acid Above a Threshold Concentration of Serum Total Folate. J Nutr. 2018 Jul 1;148(7):1103-1108. doi: 10.1093/jn/nxy070. PMID 29901753
- [Derived] March KM, Chen NN, Karakochuk CD, Shand AW, Innis SM, von Dadelszen P, Barr SI, Lyon MR, Whiting SJ, Weiler HA, Green TJ. Maternal vitamin D(3) supplementation at 50 mug/d protects against low serum 25-hydroxyvitamin D in infants at 8 wk of age: a randomized controlled trial of 3 doses of vitamin D beginning in gestation and continued in lactation. Am J Clin Nutr. 2015 Aug;102(2):402-10. doi: 10.3945/ajcn.114.106385. Epub 2015 Jul 8. PMID 26156737